CLINICAL TRIAL: NCT03895762
Title: An Observational Study to Assess the Efficacy, Safety, and Tolerability of Abstral Oral Disintegrating Tablet (ODT) for the Management of Breakthrough Cancer Pain in Korean Cancer Patients
Brief Title: Observational Study of Efficacy, Safety and Tolerability of Fentanyl in Korean Cancer Patients
Acronym: OASIS
Status: Completed | Type: Observational
Sponsor: A.Menarini Asia-Pacific Holdings Pte Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MAKR/16/Abs-Can/001
Record Dates: First submitted 2018-11-15; First posted 2019-03-29 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Breakthrough Cancer Pain
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Abstral Oral Disintegrating Tablet (ODT): Abstral Oral Disintegrating Tablet (ODT)
  Interventions: Drug: Abstral Oral Disintegrating Tablet (ODT)

INTERVENTIONS:
Drug: Abstral Oral Disintegrating Tablet (ODT) — Opioid(Fentanyl)
  Other Names: Fentanyl

SUMMARY:
The purpose of this observational study is:

To observe the efficacy, safety, and tolerability of Abstral ODT for the alleviation of breakthrough cancer pain in Korean patients with various cancers in real-world clinical settings and supplement and expand the previous cross-sectional survey results.

DETAILED DESCRIPTION:
This is a multicenter, non-interventional, single-arm, non-randomized observational study designed to collect the efficacy, safety, and tolerability data of Abstral ODT for the treatment of breakthrough cancer pain in cancer patients in real-world outpatient and inpatient clinical settings.

As the purpose of this study is to investigate the efficacy and safety of Abstral ODT in routine clinical practice, drug prescription and treatment will be determined according to the medical judgment of the investigator, regardless of enrollment to this study. During the patient's visit to the institution, Abstral ODT will be prescribed according to the judgment of the investigator, and study participation will be suggested for this patient. Whether to participate in this study or not will not affect the patient's treatment (physician's prescription or diagnostic and therapeutic decision).

Due to the non-interventional observational nature of this study, there will be no visits or procedures to be performed mandatorily according to the protocol, and data will be collected at Week 1 (±3 days), Week 4 (±1 week), and Week 12 (±4 weeks) from the baseline visit according to the circumstances of clinical practice.

Status of successful dose titration for Abstral ODT will be determined according to the criteria in which dose titration is deemed successful when all of the following are met, and ineffective when one of the following is not met: no additional dose is administered within 2 h of administration of Abstral ODT during maintenance phase; Numeric Rating Scale scores at 30 and 60 min after administration is reduced by ≥2; adverse drug reactions are tolerable for the subject.The overall procedures of this study are as follows.

ELIGIBILITY:
Inclusion Criteria:

1. Korean male and female adults at the age of 19 or older
2. In patient with Breakthrough cancer pain in inpatient or outpatient settings,

   * Patient with minimally 1 attack per day for the last week
   * Uncontrolled Breakthrough cancer pain patient with previous treatment with other fentanyl based on Invenstigator's judgment or patient who had not satisfied with previous treatment with other fentanyl at patient's request
3. Patient with opioid tolerance (treatment with at least 60 ㎎/day oral morphine, at least 25 mcg/hour transdermal fentanyl, at least 30 ㎎/day oxycodone, at least 8 ㎎/day oral hydromorphone, or other opioids at equivalent analgesic doses for 1 week or longer)
4. Patient who has been on opioids for the treatment of background cancer pain
5. Patient who did not administer Abstral ODT within 1 month prior to the baseline visit
6. Patient who signs the data release consent to data use.

Exclusion Criteria:

1. Patient for whom Abstral ODT is contraindicated based on its summary of product characteristics
2. Patient who is considered by the investigator to be ineligible for study participation for other reasons
3. Patient who is participating or participated in an opioid related clinical trial within 30 days prior to the baseline visit
4. Patient with neuropathic pain attacks

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and female patient aged 19 and over
Study Population: Patients who have been regularly on treatment with opioids for cancer pain from before study initiation and have no prior treatment with Abstral ODT within 30 days prior to study initiation.
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Number of Subjects of successful dose titration | week 1
  Status of successful dose titration. Titration is considered successful when all of the following are met, and ineffective when one of the following is not met:
  * No additional dose is administered within 2 h of administration of Abstral ODT during maintenance phase;
  * Numeric Rating Scale scores at 30 mins after administration is reduced by ≥2; Numeric Rating Scale is to measure pain intensity in subject by verbally responding to a 10-point Numeric Rating Scale (0=no pain and 10=worst possible pain in total range)
  * Adverse drug reactions are tolerable for the subject.
Number of Subjects of successful dose titration | week 4
  Status of successful dose titration. Titration is considered successful when all of the following are met, and ineffective when one of the following is not met:
  * No additional dose is administered within 2 h of administration of Abstral ODT during maintenance phase;
  * Numeric Rating Scale scores at 30 mins after administration is reduced by ≥2; Numeric Rating Scale is to measure pain intensity in subject by verbally responding to a 10-point Numeric Rating Scale (0=no pain and 10=worst possible pain in total range)
  * Adverse drug reactions are tolerable for the subject.
Number of Subjects of successful dose titration | week 12
  Status of successful dose titration. Titration is considered successful when all of the following are met, and ineffective when one of the following is not met:
  * No additional dose is administered within 2 h of administration of Abstral ODT during maintenance phase;
  * Numeric Rating Scale scores at 30 mins after administration is reduced by ≥2; Numeric Rating Scale is to measure pain intensity in subject by verbally responding to a 10-point Numeric Rating Scale (0=no pain and 10=worst possible pain in total range)
  * Adverse drug reactions are tolerable for the subject.

SECONDARY OUTCOMES:
Status of achievement of Numeric Rating Scale goal | week 1
  Status of achievement of Numeric Rating Scale goal set by each subject
  Numeric Rating Scale is to measure pain intensity in subject by verbally responding to a 10-point Numeric Rating Scale (0=no pain and 10=worst possible pain in total range)
Abstral ODT maintenance dose | week 1(dose titration)
  Abstral ODT maintenance dose at Week 4 and 12 of treatment, and after dose titration
  Data will be collected at Week 1 (±3 days), Week 4 (±1 week), and Week 12 (±4 weeks) from the baseline visit according to the circumstances of clinical practice.
Abstral ODT maintenance dose | week 4
  Abstral ODT maintenance dose at Week 4 and 12 of treatment, and after dose titration
  Data will be collected at Week 1 (±3 days), Week 4 (±1 week), and Week 12 (±4 weeks) from the baseline visit according to the circumstances of clinical practice.
Abstral ODT maintenance dose | week 12
  Abstral ODT maintenance dose at Week 4 and 12 of treatment, and after dose titration
  Data will be collected at Week 1 (±3 days), Week 4 (±1 week), and Week 12 (±4 weeks) from the baseline visit according to the circumstances of clinical practice.
Brief Pain Inventory-Korean and Pain Diary values and changes | week 1
  Brief Pain Inventory-Korean and Pain Diary values (maximum pain intensity of all incidences of breakthrough pain, pain intensity difference at 30min, pain intensity difference at 60 mins, quality of sleep, etc.) and changes. Brief Pain Inventory-Korean is to measure pain intensity in subject by verbally responding to a 10-point scale(0=no pain and 10=worst possible pain in total range)
Brief Pain Inventory-Korean and Pain Diary values and changes | week 4
  Brief Pain Inventory-Korean and Pain Diary values (maximum pain intensity of all incidences of breakthrough pain, pain intensity difference at 30min, pain intensity difference at 60 mins, quality of sleep, etc.) and changes. Brief Pain Inventory-Korean is to measure pain intensity in subject by verbally responding to a 10-point scale(0=no pain and 10=worst possible pain in total range)
Brief Pain Inventory-Korean and Pain Diary values and changes | week 12
  Brief Pain Inventory-Korean and Pain Diary values (maximum pain intensity of all incidences of breakthrough pain, pain intensity difference at 30min, pain intensity difference at 60 mins, quality of sleep, etc.) and changes. Brief Pain Inventory-Korean is to measure pain intensity in subject by verbally responding to a 10-point scale(0=no pain and 10=worst possible pain in total range)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Seok Ahn, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haugen DF, Hjermstad MJ, Hagen N, Caraceni A, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Assessment and classification of cancer breakthrough pain: a systematic literature review. Pain. 2010 Jun;149(3):476-482. doi: 10.1016/j.pain.2010.02.035. Epub 2010 Mar 16. PMID 20236762
- [Background] Davies AN, Dickman A, Reid C, Stevens AM, Zeppetella G; Science Committee of the Association for Palliative Medicine of Great Britain and Ireland. The management of cancer-related breakthrough pain: recommendations of a task group of the Science Committee of the Association for Palliative Medicine of Great Britain and Ireland. Eur J Pain. 2009 Apr;13(4):331-8. doi: 10.1016/j.ejpain.2008.06.014. Epub 2008 Aug 15. PMID 18707904
- [Background] Corli O, Floriani I, Roberto A, Montanari M, Galli F, Greco MT, Caraceni A, Kaasa S, Dragani TA, Azzarello G, Luzzani M, Cavanna L, Bandieri E, Gamucci T, Lipari G, Di Gregorio R, Valenti D, Reale C, Pavesi L, Iorno V, Crispino C, Pacchioni M, Apolone G; CERP STUDY OF PAIN GROUP (List of collaborators). Are strong opioids equally effective and safe in the treatment of chronic cancer pain? A multicenter randomized phase IV 'real life' trial on the variability of response to opioids. Ann Oncol. 2016 Jun;27(6):1107-1115. doi: 10.1093/annonc/mdw097. Epub 2016 Mar 2. PMID 26940689
- [Background] Deandrea S, Corli O, Consonni D, Villani W, Greco MT, Apolone G. Prevalence of breakthrough cancer pain: a systematic review and a pooled analysis of published literature. J Pain Symptom Manage. 2014 Jan;47(1):57-76. doi: 10.1016/j.jpainsymman.2013.02.015. Epub 2013 Jun 21. PMID 23796584
- [Background] Portenoy RK, Hagen NA. Breakthrough pain: definition, prevalence and characteristics. Pain. 1990 Jun;41(3):273-281. doi: 10.1016/0304-3959(90)90004-W. PMID 1697056
- [Background] Portenoy RK, Payne D, Jacobsen P. Breakthrough pain: characteristics and impact in patients with cancer pain. Pain. 1999 May;81(1-2):129-34. doi: 10.1016/s0304-3959(99)00006-8. PMID 10353500
- [Background] Portenoy RK, Hagen NA. Breakthrough pain: definition and management. Oncology (Williston Park). 1989 Aug;3(8 Suppl):25-9. PMID 2484297
- [Background] Zeppetella G, O'Doherty CA, Collins S. Prevalence and characteristics of breakthrough pain in cancer patients admitted to a hospice. J Pain Symptom Manage. 2000 Aug;20(2):87-92. doi: 10.1016/s0885-3924(00)00161-5. PMID 10989246
- [Background] Hong SH, Roh SY, Kim SY, Shin SW, Kim CS, Choi JH, Kim SY, Yim CY, Sohn CH, Song HS, Hong YS. Change in cancer pain management in Korea between 2001 and 2006: results of two nationwide surveys. J Pain Symptom Manage. 2011 Jan;41(1):93-103. doi: 10.1016/j.jpainsymman.2010.03.025. Epub 2010 Sep 26. PMID 20870388
- [Background] Caraceni A, Martini C, Zecca E, Portenoy RK, Ashby MA, Hawson G, Jackson KA, Lickiss N, Muirden N, Pisasale M, Moulin D, Schulz VN, Rico Pazo MA, Serrano JA, Andersen H, Henriksen HT, Mejholm I, Sjogren P, Heiskanen T, Kalso E, Pere P, Poyhia R, Vuorinen E, Tigerstedt I, Ruismaki P, Bertolino M, Larue F, Ranchere JY, Hege-Scheuing G, Bowdler I, Helbing F, Kostner E, Radbruch L, Kastrinaki K, Shah S, Vijayaram S, Sharma KS, Devi PS, Jain PN, Ramamani PV, Beny A, Brunelli C, Maltoni M, Mercadante S, Plancarte R, Schug S, Engstrand P, Ovalle AF, Wang X, Alves MF, Abrunhosa MR, Sun WZ, Zhang L, Gazizov A, Vaisman M, Rudoy S, Gomez Sancho M, Vila P, Trelis J, Chaudakshetrin P, Koh ML, Van Dongen RT, Vielvoye-Kerkmeer A, Boswell MV, Elliott T, Hargus E, Lutz L; Working Group of an IASP Task Force on Cancer Pain. Breakthrough pain characteristics and syndromes in patients with cancer pain. An international survey. Palliat Med. 2004 Apr;18(3):177-83. doi: 10.1191/0269216304pm890oa. PMID 15198130
- [Background] Boceta J, De la Torre A, Samper D, Farto M, Sanchez-de la Rosa R. Consensus and controversies in the definition, assessment, treatment and monitoring of BTcP: results of a Delphi study. Clin Transl Oncol. 2016 Nov;18(11):1088-1097. doi: 10.1007/s12094-016-1490-4. PMID 26856600
- [Background] Coluzzi PH. Cancer pain management: newer perspectives on opioids and episodic pain. Am J Hosp Palliat Care. 1998 Jan-Feb;15(1):13-22. doi: 10.1177/104990919801500105. PMID 9468974
- [Background] Patt RB, Ellison NM. Breakthrough pain in cancer patients: characteristics, prevalence, and treatment. Oncology (Williston Park). 1998 Jul;12(7):1035-46; discussion 1049-52. PMID 9684277
- [Background] Coluzzi PH, Schwartzberg L, Conroy JD, Charapata S, Gay M, Busch MA, Chavez J, Ashley J, Lebo D, McCracken M, Portenoy RK. Breakthrough cancer pain: a randomized trial comparing oral transmucosal fentanyl citrate (OTFC) and morphine sulfate immediate release (MSIR). Pain. 2001 Mar;91(1-2):123-30. doi: 10.1016/s0304-3959(00)00427-9. PMID 11240084
- [Background] Lennernas B, Hedner T, Holmberg M, Bredenberg S, Nystrom C, Lennernas H. Pharmacokinetics and tolerability of different doses of fentanyl following sublingual administration of a rapidly dissolving tablet to cancer patients: a new approach to treatment of incident pain. Br J Clin Pharmacol. 2005 Feb;59(2):249-53. doi: 10.1111/j.1365-2125.2004.02264.x. PMID 15676050
- [Background] Rauck RL, Tark M, Reyes E, Hayes TG, Bartkowiak AJ, Hassman D, Nalamachu S, Derrick R, Howell J. Efficacy and long-term tolerability of sublingual fentanyl orally disintegrating tablet in the treatment of breakthrough cancer pain. Curr Med Res Opin. 2009 Dec;25(12):2877-85. doi: 10.1185/03007990903368310. PMID 19814586
- [Background] Takigawa C, Goto F, Tanda S, Shima Y, Yomiya K, Matoba M, Adachi I, Yoshimoto T, Eguchi K. Breakthrough pain management using fentanyl buccal tablet (FBT) in combination with around-the-clock (ATC) opioids based on the efficacy and safety of FBT, and its relationship with ATC opioids: results from an open-label, multi-center study in Japanese cancer patients with detailed evaluation. Jpn J Clin Oncol. 2015 Jan;45(1):67-74. doi: 10.1093/jjco/hyu167. Epub 2014 Nov 7. PMID 25381384
- [Background] Nalamachu SR, Rauck RL, Wallace MS, Hassman D, Howell J. Successful dose finding with sublingual fentanyl tablet: combined results from 2 open-label titration studies. Pain Pract. 2012 Jul;12(6):449-56. doi: 10.1111/j.1533-2500.2011.00525.x. Epub 2012 Jan 9. PMID 22226371